CLINICAL TRIAL: NCT00842218
Title: Effect of the Severity and the Treatment (Orthosis Versus Surgery)of the Idiopathic Scoliosis on the Locomotor Mechanism of the Gait.
Brief Title: The Idiopathic Scoliosis and Its Treatment (Orthopaedic and Surgery): Effect of the Severity, the Orthosis and the Arthrodesis on the Gait
Acronym: scoliosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Banse Xavier MD, PhD, Orthopaedic Research Laboratory , Université catholique de Louvain, Brussels, Belgium
Other Study IDs: READ-Mahaudens-01
Record Dates: First submitted 2009-02-10; First posted 2009-02-12 (Estimated); Last update posted 2009-02-12 (Estimated); Status verified 2009-02

CONDITIONS: Scoliosis
Keywords: Gait; scoliosis; energy; mechanics
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purposes of this study were as follows: 1) to compare locomotion parameters (kinematic, EMG, mechanical work and energy cost changes during walking in able-bodied subjects and AIS patients,2) to evaluate the effects of the frontal curve's severity of the AIS and 3) the effects of the treatment (orthosis or surgery)on these gait parameters.

DETAILED DESCRIPTION:
Introduction X-ray studies and three-dimensional analysis in standing showed that this Adolescent Idiopathic Scoliosis was characterised by stiffness of the affected vertebral levels [3, 7, 10] with decreased segmental mobilities. The impact of this stiffness was studied during functional activity such as walking to quantify the functional dynamic consequences. During gait, thoracic AIS provided an asymmetrical trunk rotation with a lack of rotation on the convex side [8] and an excessive paravertebral muscular bilateral activity [11]. These studies included only moderate scoliosis. There were no studies approaching the effects of the severity of the scoliosis curves on gait parameters.

We hypothesize first that, the spinal deformations in AIS, producing a stiffness of the trunk, pelvic and hip motions, will deteriorate the gait by reducing the segmental mobilities, increasing the mechanical work and the energy cost and second that the severity of the frontal curves will be more damaging on this parameters. To this end, we hope to gain valuable insight as to the functional effects of the scoliosis aggravation from a more dynamic perspective.

Material Fifty-four female adolescents will be included in the study. This sample consists in two groups: healthy girls and girls with adolescent idiopathic scoliosis (divided in 3 subgroups according to the Cobb angle range) [9].

A standard full spine XRay assessment will be performed to measure the Cobb angle curve, the frontal body balance, the apical vertebral rotation [13].

Gait will be assessed by a three-dimensional analysis, including synchronous kinematic [4], electromyographic (EMG) [14], mechanic [5, 6, 15] and energetic measurements [1, 2, 12].

The sessions begins with a rest period, in which the subjects stand barefoot on the motor driven treadmill for the static calibration of kinematic and energetic variables. Thereafter, the subjects will be asked to walk at a constant speed of 4 km h-1 for a few minutes until a steady state will be reached and maintained for at least two minutes. Then, energetic variables will be computed for two minutes. Other variables will simultaneously be recorded for twenty seconds and averaged for ten successive strides. The mean of each value will be used for statistical analysis. Scoliosis patients will be assessed at T0 i.e. before any treatment and at T1 i.e. one year after the starting of the orthosis wearing (scoliosis subgroup 2) or the surgery (scoliosis subgroup 3)

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects : no scoliosis diagnosed
* Scoliosis subjects : scoliosis diagnosed by X-Ray assessment

Exclusion Criteria:

* Patients with leg length discrepancies higher than 1 cm, any locomotor disorders, low back pain, neurological abnormalities observed on clinical examination or with any previous treatment for their scoliosis

Ages: 12 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Healthy subjects girls were recruited in the town and adolescent idiopathic scoliosis attended our outpatient clinic
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-04 (Estimated); Study Completion 2009-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Mahaudens Philippe, Mr, Principal Investigator — Université Catholique de Louvain
Locations (1):
- Université Catholique de Louvain - Cliniques universitaires Saint-Luc, Brussels, Belgium

REFERENCES:
- [Background] Cavagna GA, Franzetti P, Fuchimoto T. The mechanics of walking in children. J Physiol. 1983 Oct;343:323-39. doi: 10.1113/jphysiol.1983.sp014895. PMID 6644619
- [Background] Cavagna GA, Kaneko M. Mechanical work and efficiency in level walking and running. J Physiol. 1977 Jun;268(2):467--81. doi: 10.1113/jphysiol.1977.sp011866. PMID 874922
- [Background] Danielsson AJ, Romberg K, Nachemson AL. Spinal range of motion, muscle endurance, and back pain and function at least 20 years after fusion or brace treatment for adolescent idiopathic scoliosis: a case-control study. Spine (Phila Pa 1976). 2006 Feb 1;31(3):275-83. doi: 10.1097/01.brs.0000197652.52890.71. PMID 16449899
- [Background] Davis RB OS, Tyburski D, Gage JR (1991) A gait analysis data collection and reduction technique. Hum Mov Sci 10:575-587
- [Background] Detrembleur C, van den Hecke A, Dierick F. Motion of the body centre of gravity as a summary indicator of the mechanics of human pathological gait. Gait Posture. 2000 Dec;12(3):243-50. doi: 10.1016/s0966-6362(00)00081-3. PMID 11154935
- [Background] Detrembleur C, Vanmarsenille JM, De Cuyper F, Dierick F. Relationship between energy cost, gait speed, vertical displacement of centre of body mass and efficiency of pendulum-like mechanism in unilateral amputee gait. Gait Posture. 2005 Apr;21(3):333-40. doi: 10.1016/j.gaitpost.2004.04.005. PMID 15760750
- [Background] Karski T. Biomechanical factors in the etiology of idiopathic scoliosis: two etiopathological groups of spinal deformities. Ortop Traumatol Rehabil. 2004 Nov-Dec;6(6):800-8. PMID 17618198
- [Background] Kramers-de Quervain IA, Muller R, Stacoff A, Grob D, Stussi E. Gait analysis in patients with idiopathic scoliosis. Eur Spine J. 2004 Aug;13(5):449-56. doi: 10.1007/s00586-003-0588-x. Epub 2004 Apr 3. PMID 15064994
- [Background] Lenke LG, Betz RR, Harms J, Bridwell KH, Clements DH, Lowe TG, Blanke K. Adolescent idiopathic scoliosis: a new classification to determine extent of spinal arthrodesis. J Bone Joint Surg Am. 2001 Aug;83(8):1169-81. PMID 11507125
- [Background] Leong JC, Lu WW, Luk KD, Karlberg EM. Kinematics of the chest cage and spine during breathing in healthy individuals and in patients with adolescent idiopathic scoliosis. Spine (Phila Pa 1976). 1999 Jul 1;24(13):1310-5. doi: 10.1097/00007632-199907010-00007. PMID 10404572
- [Background] Mahaudens P, Thonnard JL, Detrembleur C. Influence of structural pelvic disorders during standing and walking in adolescents with idiopathic scoliosis. Spine J. 2005 Jul-Aug;5(4):427-33. doi: 10.1016/j.spinee.2004.11.014. PMID 15996612
- [Background] McArdle W, Katch F, Katch V (1996) Exercise physiology: Energy, Nutrition, and Human Performance. Baltimore
- [Background] Roche AF, Eyman SL, Davila GH. Skeletal age prediction. J Pediatr. 1971 Jun;78(6):997-1003. doi: 10.1016/s0022-3476(71)80430-4. No abstract available. PMID 4325224
- [Background] Van Boxtel GJ, Geraats LH, Van den Berg-Lenssen MM, Brunia CH. Detection of EMG onset in ERP research. Psychophysiology. 1993 Jul;30(4):405-12. doi: 10.1111/j.1469-8986.1993.tb02062.x. PMID 8327626
- [Background] Willems PA, Cavagna GA, Heglund NC. External, internal and total work in human locomotion. J Exp Biol. 1995 Feb;198(Pt 2):379-93. doi: 10.1242/jeb.198.2.379. PMID 7699313